CLINICAL TRIAL: NCT05089968
Title: Ventilator-associated Pneumonia Ecology Comparison in a French ICU Center NIMES Between First and Second Wave of COVID-19 : a Retrospective Monocentric Descriptive Study
Brief Title: Ventilation Associated Pneumonia and Covid-19
Acronym: ECOLCOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/LC-01
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV2 Infection; Ventilator Associated Pneumonia; Ards; COVID-19
Keywords: Intensive care Unit; multidrug resistance; COVID 19 ARDS; ventilator associated pneumonia; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19; Pneumonia, Ventilator-Associated; Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient from the first wave of COVID-19: 57 Patients hospitalized in intensive care unit for pneumonia related to a Sars-Cov2 infection who required mechanical ventilatory support and developed microbiologically documented ventilator associated pneumonia during the 1st wave from January 24, 2020 to July 10, 2020
- Patient from the Second wave of COVID-19: 211 Patients hospitalized in intensive care unit for pneumonia related to a Sars-Cov2 infection who required mechanical ventilatory support and developed microbiologically documented ventilator associated pneumonia during the 2nd wave from July 11, 2020 to January 8, 2021

SUMMARY:
In December 2019, a new pandemic emerged, the COVID-19 disease caused by a SARS-Cov-2 virus. One of the most common symptoms of COVID-19 is mainly respiratory failure and patients requires assistance by mechanical ventilation. Ventilator-associated pneumonia (VAP) is a risk of this assistance. Since the beginning of the pandemic, Standard of care have evolved with new data. The prevalence of these VAPs seems significantly higher in the population of patients with ARDS COVID-19 (40-50%) and their ecology seems to have evolved over time, particularly in terms of bacterial resistance. Investigators want to describe and compare this evolution of bacterial and fungal ecology as well as identify potential risk factors that may be associated with these changes in ecology during different waves.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Positive SARS-Cov-2 polymerase chain reaction (PCR)
* healthcare associated pneumonia

Exclusion Criteria : Patient opposition to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with a SARS-CoV-2 infection confirmed by positive PCR tests of nasopharyngeal or respiratory secretion samples. In addition, patients included presented a healthcare associated pneumonia according to SFAR(French Society of Anesthesia and Intensive Care) recommendations and based on criteria adapted from the European Centre for Disease Prevention and Control (ECDC) recommendations. Patients who refused their data use were excluded.
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
VAP ecological difference between the first and second waves of COVID | January 2020 to January 2021
  Proportion of patients admitted to critical care with documented multidrug-resistant bacteria (MDR) VAP in Covid-19 wave 1 and 2

SECONDARY OUTCOMES:
proportion of fungal co-infections | January 2020 to January 2021
  Comparison of the proportion of patients with a fungal infection during the 1st and 2nd wave
duration of mechanical ventilation | Day 28
  Number of days under mechanical ventilations
number of days of organ failure | Day 28
  number of days between first organ failure and no organ failure (discharge from intensive care)
Mortality | Day 28
  proportion of patients deceased at day 28
proportion of patients treated with corticosteroid therapy | Day 28
  proportion of patients treated with corticosteroid therapy
probabilistic antibiotic therapy at admission | Day 1
  probabilistic antibiotic therapy prescribed at admission
antiviral treatment | Day 28
  proportion of patients treated with antiviral treatment

CONTACTS AND LOCATIONS:
Overall Officials: Claire ROGER, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No